CLINICAL TRIAL: NCT06987864
Title: An Extension Clinical Study of BCD-148 (JSC BIOCAD) for the Treatment of Patients With Paroxysmal Nocturnal Hemoglobinuria Previously Treated in Clinical Study No. BCD-148-2/NOCTURN
Brief Title: An Extension Clinical Study of BCD-148 for the Treatment of Patients With PNH Previously Treated in Clinical Study No. BCD-148-2/NOCTURN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCD-148-EXT
Record Dates: First submitted 2025-05-16; First posted 2025-05-23 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria (PNH)
Keywords: Paroxysmal nocturnal hemoglobinuria; eculizumab; PNH
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal | interventions — eculizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- To study the long-term safety and efficacy of BCD-148 in patients with paroxysmal nocturnal hemoglob (Experimental)
  Interventions: Biological: eculizumab

INTERVENTIONS:
Biological: eculizumab — Intravenous infusion of BCD-148 every 2 weeks

SUMMARY:
To study the long-term safety and efficacy of BCD-148 in patients with paroxysmal nocturnal hemoglobinuria (PNH), previously treated in clinical study (CS) BCD-148-2/NOCTURN

DETAILED DESCRIPTION:
The clinical study BCD-148-EXT was an extension of a multicenter, randomized, open-label, comparative study of the efficacy and safety of BCD-148 in PNH patients versus SOLIRIS® (BCD-148-2/NOCTURN).

Clinical study BCD-148-EXT is a Phase III study extension conducted after completion of BCD-148 900 mg therapy or SOLIRIS® 900 mg by subjects of clinical study BCD-148-2/NOCTURN.

In the BCD-148-EXT clinical study patients continued BCD-148 maintenance therapy for 105 weeks.

The BCD-148-EXT study consisted of two periods: screening period (not more than 7 days inclusive, i.e. 1 week from signing the patient information sheet and IC form) and the treatment period (Weeks 0 to 105 of the study, inclusive). As part of the treatment period, patients received intravenous infusions of the investigational drug BCD-148 in the maintenance therapy regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Signed IC form for participation in the study.
2. Indications for pathogenesis-based therapy of PNH with an anti-C5 monoclonal antibody (eculizumab).
3. Consent for revaccination against Neisseria meningitidis .
4. Negative pregnancy test for urine human chorionic gonadotropin (HCG) in women at enrollment in study BCD-148-EXT (the test was not performed in women who have been postmenopausal for at least 2 years, or in surgically sterile subjects) .
5. Willingness of patients and their sexual partners of childbearing potential to use reliable contraceptive measures from signing the IC form throughout the study and for 4 weeks after the last drug dosing in the clinical study. This requirement did not apply to patients who underwent surgical sterilization and women who have been postmenopausal for over 2 years. Reliable methods of contraception included the use by partners of one barrier method in combination with one of the following: spermicides, intrauterine device, oral contraceptives (for female partners of male subjects only, for female study participants - upon agreement with the Sponsor and with justification by the investigator) .
6. The ability of the patient to comply with the Protocol requirements, in the Investigator's opinion.

Exclusion Criteria:

1. Patient withdrawal from clinical study BCD-148-2/NOCTURN until its completion for any reason.
2. Pregnancy or breastfeeding, or planning of pregnancy by a female participant/planning conceiving a child by a male participant during the clinical study.
3. Any conditions that, in the investigator's opinion, could increase the patient's risk associated with participation in the study or could affect the assessment of the study results.
4. Hypersensitivity to BCD-148 components, murine proteins, and other components of the products according to the patient's history; hypersensitivity to any component of the meningococcal vaccine.
5. Known alcohol or drug addiction, or signs of alcohol/drug addiction, which, according to the investigator, were a contraindication for the treatment with the study drug or limited the treatment compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-04-13 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2022-11-02 (Actual)

PRIMARY OUTCOMES:
Change in lactate dehydrogenase (LDH) level from baseline estimated at Visit 1/Week 0 prior to drug administration | 105 weeks

SECONDARY OUTCOMES:
Proportion of patients with thrombotic complications | 105 weeks
Change in the size of the PNH clone (change in the number of circulating red blood cells with the PNH phenotype) from baseline estimated at Visit 1/Week 0 prior to drug administration | 105 weeks
Change in the mean Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Scale Total Score from baseline as assessed at Visit 1/Week 0 prior to drug administration | 105 weeks
  The assessment of the quality of life of patients was carried out on the basis of the analysis of change in the mean score on the FACIT-Fatigue scale at Visits 1-14 (Weeks 0-104) compared to the baseline values. An increase in the score indicates a decrease in the patient's fatigue severity.
Proportion of patients with adverse reactions (ARs), including those meeting the seriousness criteria | 105 weeks
Proportion of patients with grade 3 or higher adverse reactions (ARs) according to the Common Toxicity Criteria for Adverse Events (CTCAE) version 5.0 | 105 weeks
  Proportion of patients with grade 3, 4 or 5 ARs according to the CTCAE v.5.0
Proportion of patients who prematurely withdrew from the study due to ARs | 105 weeks
Proportion of BAb (binding antibodies) and NAb (neutralizing antibodies)-positive patients | 105 weeks
Eculizumab Ctrough (steady-state eculizumab concentration at the end of the dosing interval, before the next scheduled dose, after multiple intravenous infusions of BCD-148) | 105 weeks
Emin of serum complement hemolytic activity and C5 level (minimum serum complement hemolytic activity and C5 levels after administration of BCD-148) | 105 weeks
Etrough of serum complement hemolytic activity and C5 level (the effect magnitude measured at the end of the dosing interval, before the next scheduled dose, at steady state after multiple intravenous infusions of BCD-148) | 105 weeks

CONTACTS AND LOCATIONS:
Locations (11):
- Russia (11):
  - Territorial State Budgetary Healthcare Institution "Territorial Clinical Hospital", Barnaul
  - State Autonomous Healthcare Institution "S.V. Belyaev Kuzbass Regional Clinical Hospital", Kemerovo
  - Federal State Budgetary Institution of Science "Kirov Research Institute of Hematology and Blood Transfusion of the Federal Medical and Biological Agency", Kirov
  - Moscow State Budgetary Healthcare Institution "S.P. Botkin Municipal Clinical Hospital of the Moscow Healthcare Department", Moscow
  - Federal State Budgetary Educational Institution of Higher Education "Rostov State Medical University" of the Ministry of Health of the Russian Federation, Rostov-on-Don
  - Federal State Budgetary Educational Institution of Higher Education "Academician I.P. Pavlov First St. Petersburg State Medical University" of the Ministry of Health of the Russian Federation, Saint Petersburg
  - Federal State Budgetary Educational Institution of Higher Education "I.I. Mechnikov North-Western State Medical University" of the Ministry of Health of the Russian Federation, Saint Petersburg
  - Federal State Budgetary Educational Institution of Higher Education "Samara State Medical University" of the Ministry of Health of the Russian Federation, Samara
  - State Institution "Komi Republican Cancer Clinic", Syktyvkar
  - Federal State Budgetary Educational Institution of Higher Education "Bashkir State Medical University" of the Ministry of Health of the Russian Federation, Ufa
  - State Autonomous Healthcare Institution of the Sverdlovsk Region "Sverdlovsk Regional Clinical Hospital No. 1", Yekaterinburg